CLINICAL TRIAL: NCT06210009
Title: Effect of a DASH-Style Diet on Urinary Risk Factors for Kidney Stone Disease: A Randomized Controlled Trial (CARDIA Ancillary Study)
Brief Title: Effect of a DASH-Style Diet on Urinary Risk Factors for Kidney Stone Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Joseph Crivelli, Assistant Professor of Urology, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB-300012217
Record Dates: First submitted 2024-01-04; First posted 2024-01-18 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Kidney Stone
Keywords: DASH diet; Western diet
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DASH-Style Diet (Experimental): For seven days, participants will consume a diet characterized by higher intake of fruits, vegetables, and low-fat dairy, in addition to whole grains, poultry, fish, and nuts, but smaller amounts of red meat, sweets, and sugar-containing beverages.
  Interventions: Other: DASH-Style Diet
- Western-Style Diet (Other): For seven days, participants will consume a diet characterized by characterized by higher intake of red meat, sweets, and items containing added sugar, processed starches, and seed oils, in addition to lower intake of fruits, vegetables, and low-fat dairy.
  Interventions: Other: Western-Style Diet

INTERVENTIONS:
Other: DASH-Style Diet — Participants will be randomized to a DASH-style diet
  Arms: DASH-Style Diet
Other: Western-Style Diet — Participants will be randomized to a Western-style diet
  Arms: Western-Style Diet

SUMMARY:
The true capacity for a healthy diet to improve urinary stone risk factors is not well-defined. The objective of this study is to measure the effect of adopting a healthy dietary pattern on kidney stone disease (KSD) risk. The working hypothesis is that a Dietary Approaches to Stop Hypertension (DASH)-style diet will improve 24-hour urine stone risk parameters. The approach to testing this hypothesis will be to randomize participants with KSD to a standardized DASH-style vs. Western-style diet for one week. The Bionutrition Unit of the Center for Clinical and Translational Science will provide all meals to participants. The rationale for this study is that by measuring the effect of a DASH-style diet on urinary stone risk parameters, a benchmark for future real-world, implementation studies will be established. Based on available evidence, this will be the first controlled diet study to assess the DASH dietary pattern for improving urinary stone risk parameters.

ELIGIBILITY:
Inclusion Criteria:

* Birmingham, AL area participants of the Coronary Artery Risk Development in Young Adults (CARDIA) study OR patients of the University of Alabama at Birmingham/Kirklin Clinic
* Self-reported, documented, and/or prior imaging-based diagnosis of kidney stone disease
* Age 19-89
* Any sex
* Any race
* Able to provide informed consent
* Willing to perform 24-hour urine collections
* Willing to consume meals prepared by Bionutrition Unit
* No food allergies/intolerance to any of the foods in the study menus
* Willing to stop for 7 days before and during study: Multivitamins and/or Dietary supplements (including calcium and vitamin C)

Exclusion Criteria:

* Dialysis
* Kidney transplant recipient
* Estimated glomerular filtration rate (eGFR) <60 ml/min/1.73m2 based on historical laboratory measurements
* Renal tubular acidosis
* Current use of acetazolamide, topiramate, or zonisamide
* Primary hyperparathyroidism or history of parathyroidectomy
* Hyperthyroidism
* Sarcoidosis
* Primary hyperoxaluria
* Cystinuria
* Nephrotic syndrome
* Malabsorptive conditions including inflammatory bowel disease or history of malabsorptive surgery (e.g., Roux-en-Y gastric bypass, small bowel resection)
* Urinary retention requiring catheterization
* Urinary diversion
* Pregnancy
* Breastfeeding
* Malignancy treated in the past 12 months other than non-melanoma skin cancer

Ages: 19 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Difference between the two arms in supersaturation of calcium oxalate | Days 6-7 of the assigned intervention
  Supersaturation of calcium oxalate is an index reflecting the propensity for the formation and growth of the most common stone type (calcium oxalate), which is calculated using excretion rates including urinary volume, calcium, citrate, and oxalate.

SECONDARY OUTCOMES:
Difference between the two arms in supersaturation of calcium oxalate between the baseline and intervention periods | Days 6-7 of the assigned intervention
  This secondary outcome will be calculated using a difference in differences approach.
Difference between the two arms in supersaturation of uric acid | Days 6-7 of the assigned intervention
  Supersaturation of uric acid is an index reflecting the propensity for the formation and growth of uric acid stones.
Difference between the two arms in supersaturation of calcium phosphate | Days 6-7 of the assigned intervention
  Supersaturation of calcium phosphate is an index reflecting the propensity for the formation and growth of calcium phosphate stones.
Difference between the two arms in urine volume | Days 6-7 of the assigned intervention
  Low urine volume is a stone risk factor.
Difference between the two arms in urine calcium | Days 6-7 of the assigned intervention
  High urine calcium is a stone risk factor.
Difference between the two arms in urine oxalate | Days 6-7 of the assigned intervention
  High urine oxalate is a stone risk factor.
Difference between the two arms in urine citrate | Days 6-7 of the assigned intervention
  Low urine citrate is a stone risk factor.
Difference between the two arms in urine uric acid | Days 6-7 of the assigned intervention
  High urine uric acid is a stone risk factor.
Difference between the two arms in urine pH | Days 6-7 of the assigned intervention
  Urine pH can influence stone formation and growth.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States